CLINICAL TRIAL: NCT03318445
Title: Combination Therapy of Rucaparib and Irinotecan in Cancers With Mutations in DNA Repair
Brief Title: Rucaparib and Irinotecan in Cancers With Mutations in DNA Repair
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pamela Munster (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Pamela Munster, Professor, Department of Medicine; Director, Early Phase Clinical Trials Unit, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 169521; NCI-2017-02294 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor, Unspecified, Adult
Keywords: DNA repair mutation
MeSH Terms: interventions — rucaparib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rucaparib and irinotecan (Experimental): Rucaparib will be taken twice daily by mouth for 7-14 days in 21 or 28 day cycles. Irinotecan will be administered by IV for 90 minutes every 14 days, or every 21 days if not tolerated.
  During the dose escalation phase, the maximum tolerated dose for combining Rucaparib and irinotecan will be determined. The dose for rucaparib during dose escalation will range from 300 mg to 600 mg, depending on the progression of study. The dose for irinotecan during dose escalation may range from 40 mg/m2 to 150 mg/m2.
  During the dose expansion phase, patients who have received prior PARP inhibitors will be given rucaparib and irinotecan at the maximum tolerated dose levels determined during the dose escalation phase.
  Interventions: Drug: Rucaparib; Drug: Irinotecan
- Rucaparib only (Experimental): During the dose expansion phase, patients who have not received prior PARP inhibitor therapy will take 600 mg of rucaparib by mouth daily. Patients who progress on single-agent rucaparib will be given the option to cross-over to the combination treatment arm and receive rucaparib in combination with irinotecan at the maximum tolerated dose levels determined during dose escalation.
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — All participants will take rucaparib by mouth
  Other Names: Rubraca
Drug: Irinotecan — Patients in the dose escalation phase, and patients in the dose expansion phase who have received prior PARP inhibitor therapy, will be given irinotecan by in combination with rucaparib.
  Other Names: Camptosar
  Arms: Rucaparib and irinotecan

SUMMARY:
This is an open label, non-randomized, dose escalation and expansion Phase Ib trial to evaluate the safety and recommended phase II dose of the combination of irinotecan and rucaparib.

DETAILED DESCRIPTION:
In dose escalation, patients will receive irinotecan and rucaparib. Irinotecan will be given once every 2 weeks (or 3 weeks if not tolerated) and rucaparib will be given twice daily for 7-14 days. Each cycle will be 28 days in duration unless we need to switch to the intermediate dosing regimen of every 21 days. Both rucaparib and irinotecan will be escalated.

In dose expansion, patients who have received prior PARP inhibitors will go straight to the combination arm of irinotecan and rucaparib. If patients are PARP inhibitor naïve, they can receive single agent rucaparib until progression. Once patients on single agent rucaparib progress, they can choose to go on the combination treatment arm. Patients will continue on treatment until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria for Dose Escalation Cohort:

1. Men and women, 18 years or older
2. Understand and voluntarily sign informed consent prior to any study-related assessments or procedures are conducted and are able adhere to the study visit schedule and other protocol requirements.
3. Solid tumors with one or more of the following DNA repair defects:

   a. BRCA1, BRCA2, ATM, BARD1, BRIP1, CDK12, CHEK2, FANCA, NBN, PALB2, RAD51, RAD51B, RAD51C, RAD51D, RAD54L (validated from archival tumor tissue or germ line testing from any Clinical Laboratory Improvement Amendments (CLIA) approved lab). This testing should occur prior to study consent or enrollment.
4. Presence of at least one lesion with measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria for response assessment
5. Advanced solid tumor malignancy without curative options
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1.
7. Adequate organ function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 X 109/L
   2. Hemoglobin (Hgb) ≥9g/dL; (last transfusion cannot be within 7 days of trial initiation)
   3. Platelets (plt) ≥ 100 x 109/L
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x Upper Limit Normal (ULN), <5x in patients with known liver metastases
   5. Serum total bilirubin ≤ 1.5 x ULN
   6. Creatinine<1.5 x ULN or estimated Glomerular filtration rate (GFR) ≥ 50ml/min by Cockcroft-Gault (http://www.mdcalc.com/creatinine-clearance-cockcroft-gault-equation/)
8. The effects of rucaparib on the developing fetus are unknown. Therefore a. Given the results of the embryo-fetal development study, in which rucaparib was embryotoxic at all doses administered, females of childbearing potential and their male partners are advised to practice a highly effective method of contraception during treatment with rucaparib and for 1 month following the last dose for females and 4 months following the last dose for males. A woman is considered to be of childbearing potential unless one of the following applies: i. Is considered to be permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   ii. Is postmenopausal, defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level consistently in the postmenopausal range (30 milli-international units per millilitre (mIU/mL) or higher) may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to confirm a postmenopausal state.

   b. Highly effective contraception is considered to be a method with a < 1% per year failure rate. Recommendations for highly effective contraception while taking rucaparib include: i. Ongoing use of injectable or implantable progesterone ii. Placement of an intrauterine device or intrauterine system iii. Bilateral tubal occlusion iv. Complete (as opposed to periodic) abstinence v. Male sterilization, with appropriate post-vasectomy documentation of absence of sperm in ejaculate

   Additional Inclusion Criteria for Dose Expansion Cohort
9. Mandatory biopsy on study entry, if the lesion can be biopsied with acceptable clinical risk (as judged by the investigator)
10. PARP inhibitor (PARPi) naïve or prior exposure to PARPi therapy (varies depending on Arm 1 and Arm 2)

    1. Patients in Arm 1 (single agent rucaparib followed by combination upon progression) must be PARPi naïve. Prior irinotecan is allowed
    2. Patients in Arm 2 (combination) must have been treated with and progressed on a PARPi previously. Prior irinotecan is allowed.

Exclusion Criteria for Dose Escalation Cohort:

1. Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study at clinician's discretion and not otherwise stated below.
2. Allergic reaction to single-agent rucaparib or irinotecan.
3. Myelodysplastic features on peripheral blood smear
4. Prior allergic reaction or known intolerance to irinotecan
5. Known Gilbert's disease
6. Poorly controlled or symptomatic central nervous system (CNS) metastases or carcinomatous meningitis

Note: Patients with previously treated brain metastases may participate, 2 weeks after gamma knife (or equivalent) or 4 weeks after Whole Brain Radiotherapy (WBRT), provided they are stable (without evidence of progression by imaging and have not been using steroids for at least 7 days prior to study treatment.

8. Pregnancy and breast feeding

9. Inability to comply with study procedures or willingness to use adequate birth control

Additional Exclusion Criteria for Dose Expansion Cohort

10. PARP inhibitors (PARPi) naïve or prior exposure to PARPi therapy

1. Patients in Arm 1 of the Dose Expansion cohort cannot have prior exposure to PARPi therapy.
2. Patients in Arm 2 of the Dose Expansion cohort cannot be PARPi naïve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months.
  ORR is defined as the proportion of patients with either confirmed complete or partial response (as per RECIST version 1.1) as best overall response over the total population.

SECONDARY OUTCOMES:
Median Response duration | Up to 24 months
  Response duration is defined as the time from initial response to the first documented tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No